CLINICAL TRIAL: NCT03529383
Title: Randomized Controlled Trial Evaluating the Efficacy of an Adapted Physical Activity Program Using a Connected Device With Activity Trackers and a Therapeutic Education Program Among Women With Localized Breast Cancer
Brief Title: Efficacy of Exercise Using Connected Activity Trackers and Therapeutic Education in Localized Breast Cancer
Acronym: DISCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: Fondation ARC (Other); National Cancer Institute, France (Other Government); Fondation pour la Recherche Médicale (Other); Cancéropôle Lyon Auvergne Rhône-Alpes (Other); AG2R La Mondiale (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: ET17-203 DISCO
Record Dates: First submitted 2018-04-13; First posted 2018-05-18 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Localized breast cancer; Exercise; Adapted physical activity; Sedentary; Connected device; Activity trackers; Therapeutic education; Obesity
MeSH Terms: conditions — Breast Neoplasms; Motor Activity; Sedentary Behavior; Obesity

STUDY DESIGN:
Intervention Model Description: Two interventions, each alone and in combination, are evaluated in parallel against a control group. Women assigned to the "connected device" arm will follow a 6-month exercise program using a connected device. Women assigned to the "therapeutic education" arm will follow a 6-month program of therapeutic patient education in physical activity. Women assigned to the "combined" arm will follow both programs. Women assigned to the "control" arm will receive international recommendations on physical activity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Connected device (Experimental): Women randomized to the "connected device" arm will follow a 6-month exercise program using a connected device that includes an activity tracker and subscription to an exercise and physical activity management program through a smartphone application and a website. They will also receive international recommendations on physical activity.
  Interventions: Device: Connected device
- Therapeutic education (Experimental): Women randomized to the "therapeutic education" arm will follow a 6-month program of therapeutic patient education. They will also receive international recommendations on physical activity.
  Interventions: Behavioral: Therapeutic education
- Combined (Experimental): Women will benefit from both the "connected device" intervention and the "therapeutic education" intervention and receive international recommendations on physical activity.
  Interventions: Device: Connected device; Behavioral: Therapeutic education
- Control (No Intervention): Women will receive standard care, i.e., international recommendations on physical activity, without further intervention.

INTERVENTIONS:
Device: Connected device — Women will receive a connected wristband (https://www.carefitness.com/) and a subscription to a smartphone application and website (http://disco.biomouv.com/). They will have to participate in a 6-month personalized non-supervised exercise program consisting of 3 weekly sessions of 20 min to 1-hr of moderate-to-vigorous physical activity (≥3 METs): 2 sessions of brisk walking and 1 session of muscle strengthening. Women should wear the wristband daily to track their number of steps (automatic Bluetooth synchronization to the application). Duration and intensity of sessions and target number of daily steps will progressively increase (+15% up to 10,000 steps) to place the patients in a progression dynamic. Women will receive phone-based follow-up at 1 week, 2 months, and 4 months.
  Arms: Combined; Connected device
Behavioral: Therapeutic education — Women will be invited to participate in the 6-month therapeutic patient education program "Mieux manger, mieux bouger" ("Eat better, move better") elaborated at the Léon Bérard cancer center. The program consists in four sessions:
  * a 1-hour individual session of "educational diagnosis" to assess their needs and establish a contract of objectives,
  * two "educational sessions" of 1h30 each using tools, in group of 10 patients maximum to improve their daily practice of physical activity,
  * a 1-hour individual session of "educational assessment" to evaluate whether their objectives were reached.
  Arms: Combined; Therapeutic education

SUMMARY:
The 3-year DISCO study aims to systematically implement physical activity in breast cancer patients. The primary objective is to investigate the efficacy of a connected device (personalized non-supervised exercise program including a wristband as activity tracker, a smartphone application, and a website) and the efficacy of a therapeutic education program on the physical activity level of patients at the end of the 6-month programs. The research hypothesis is that patients participating in the intervention with the connected device or in the therapeutic education program will achieve the international recommendations in terms of physical activity, compared to women receiving only physical activity recommendations.

DETAILED DESCRIPTION:
Rationale:

In women with breast cancer, weight gain, obesity, and lack of physical activity have been shown to increase the risk of comorbidities and deleterious long-term outcomes. Despite the safety of physical activity and the benefits of physical activity performed concomitant to treatment on fatigue, quality of life, and possibly survival, its implementation is not systematic in the cancer care pathway.

Methods:

The DISCO study is a randomized, controlled, multicenter intervention study that will be conducted among 432 women treated for localized breast cancer. Patients will be randomly assigned to one of the four arms of the study according to a 1:1:1:1 ratio.

* Women allocated to the "connected device" arm will benefit from a 6-month personalized exercise program consisting of three weekly sessions of aerobic and strength exercises, carried out autonomously with a connected device (wristband, smartphone application, website).
* Women allocated to the "therapeutic education" arm will follow a 6-month program of therapeutic patient education.
* Women allocated to the "combined" arm will benefit from both interventions in parallel.
* Women allocated to the "control" arm will receive standard care, i.e., international recommendations on physical activity.

Evaluations will be conducted at inclusion (T1, baseline), 6 months (T2, end of interventions), and 12 months (T3, 12 months post-inclusion to study maintenance of behavior change) on the following parameters: level of physical activity and sedentary behavior (RPAQ self-administered questionnaire), physical condition assessed by functional tests (6-min walking test, sit-to-stand test, hang-grip test, sit-and-reach flexibility test, single-leg balance test), anthropometrics (weight, height, waist circumference, hip circumference, calculated body mass index), body composition (fat mass, lean body mass, fat free mass, water), biological factors (blood sample at baseline and 6 months), lifestyle factors (tobacco status, alcohol intake), psychological factors (quality of life assessed by the EORTC QLQ-C30 / BR-23 questionnaire, health-related quality of life assessed by the EQ-5D-5L questionnaire, fatigue assessed by the PFS-12 questionnaire), socio-economic parameters (social deprivation assessed by the EPICES questionnaire, level of education, family situation, professional status assessed through a self-administered questionnaire). Clinical data will be obtained from patients' medical records. Acceptability of connected device and of therapeutic education program will be assessed within the population. The medico-economic impact of the interventions will be evaluated through cost-utility and cost-effectiveness analyses. Data will be recorded using an e-CRF. Women will be recruited over 2 years and will be followed up for 12 months.

Hypothesis:

The research hypothesis is that patients participating in the 6-month intervention with the connected device or in the 6-month therapeutic education program will be more likely to achieve the international recommendations in terms of physical activity, compared to women receiving only physical activity recommendations.

Expected results are to identify best modalities to implement exercise during and after breast cancer treatment. In a public health perspective, the challenge is to reduce geographical, social, and organizational inequalities among patients to practice regular physical activity and to promote the systematic integration of physical activity in routine cancer care.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 75 years old,
* Being diagnosed with a first primary non-metastatic invasive breast carcinoma, that has been histologically conﬁrmed,
* Having been operated and requiring the prescription of an adjuvant treatment (chemotherapy, hormonotherapy, radiotherapy),
* Whose adjuvant treatment will be prescribed (for hormone therapy) or carried out (for chemotherapy and radiotherapy) in one of the investigating centers,
* Being able to practice adapted physical activity and providing a medical certiﬁcate of no contraindications to exercise issued by the investigator physician, the general practitioner, or the referring physician,
* Available and willing to participate in the study for the duration of the interventions and follow-up,
* Using a personal smartphone compatible with the application (iOS operating system from version 9.3, Android operating system from version 5.0, no Microsoft operating system) and having Internet access on a computer,
* Able to understand, read, and write French,
* Affiliated with a social security scheme,
* Having dated and signed an informed consent.

Exclusion Criteria:

* Woman with recurrent, metastatic, or inflammatory breast cancer,
* Personal history or co-existence of another primary cancer (except of in situ cancer regardless of the site and/or basal cell skin cancer and/or non-mammary cancer in complete remission for more than 5 years),
* Presenting a contraindication to exercise according to the investigator (such as cardiorespiratory or bone pathologies, non-stabilized chronic diseases such as diabetes, malnutrition, etc.),
* In a state of severe malnutrition according to the criteria of the French National Health Authority (i.e., in women ≤ 70 years: weight loss ≥ 15% in 6 months or ≥ 10% in 1 month; in women > 70 years: weight loss ≥ 15% in 6 months or ≥ 10% in 1 month, and body mass index < 18 kg/m²),
* Unable to be followed for medical, social, family, geographic or psychological reasons for the duration of the study,
* Participating in simultaneous physical activity studies,
* Deprived of their liberty by court or administrative decision,
* Pregnant or breastfeeding or of childbearing age without effective contraception for the duration of the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 436 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2022-03-04 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Number of patients achieving the internationally recommended level of physical activity of at least 150 minutes per week of moderate-to-vigorous physical activity (intensity ≥3 METs) | 6 months
  Assessed by the RPAQ self-administered questionnaire

SECONDARY OUTCOMES:
Number of patients achieving the internationally recommended level of physical activity of at least 150 minutes per week of moderate-to-vigorous physical activity (intensity ≥3 METs) | 12 months
  Assessed by the RPAQ self-administered questionnaire
Proportion of patients who are compliant to the programs | 6 months
  Participation rate in planned sessions
Proportion of patients who change their physical activity profile (Time spent in different intensities of physical activity, time spent in sedentary activities) | Change between baseline and 6 months and between 6 months and 12 months
  Time spent in different intensities of physical activity, time spent in sedentary activities
Proportion of patients who change their physical condition (6-min walking test) | Change between baseline and 6 months and between 6 months and 12 months
  6-min walking test
Proportion of patients who change their physical condition (Sit to stand test) | Change between baseline and 6 months and between 6 months and 12 months
  Sit to stand test
Proportion of patients who change their physical condition (Hand-grip test) | Change between baseline and 6 months and between 6 months and 12 months
  Hand-grip test
Proportion of patients who change their physical condition (sit-and-reach flexibility test) | Change between baseline and 6 months and between 6 months and 12 months
  sit-and-reach flexibility test
Proportion of patients who change their physical condition | Change between baseline and 6 months and between 6 months and 12 months
  single-leg balance test
Proportion of patients who change their weight | Change between baseline and 6 months and between 6 months and 12 months
  Weight in kilograms
Proportion of patients who change their waist circumference | Change between baseline and 6 months and between 6 months and 12 months
  Waist circumference in cms
Proportion of patients who change their hip circumference | Change between baseline and 6 months and between 6 months and 12 months
  Hip circumference in cms
Proportion of patients who change their BMI | Change between baseline and 6 months and between 6 months and 12 months
  weight in kilograms and height in meters will be combined to report BMI in kg/m^2
Proportion of patients who change their fat mass in body composition | Change between baseline and 6 months and between 6 months and 12 months
  fat mass measured using bioelectronic impedancemetry
Proportion of patients who change their lean body mass in body composition | Change between baseline and 6 months and between 6 months and 12 months
  lean body mass measured using bioelectronic impedancemetry
Proportion of patients who change their fat free mass in body composition | Change between baseline and 6 months and between 6 months and 12 months
  fat free mass measured using bioelectronic impedancemetry
Proportion of patients who change their water in body composition | Change between baseline and 6 months and between 6 months and 12 months
  water measured using bioelectronic impedancemetry
Proportion of patients who change their tobacco use | Change between baseline and 6 months and between 6 months and 12 months
  Self-administered questionnaire
Proportion of patients who change their alcohol intake | Change between baseline and 6 months and between 6 months and 12 months
  Self-administered questionnaire
Proportion of patients with a change in quality of life | Change between baseline and 6 months and between 6 months and 12 months
  EORTC QLQ-C30 questionnaire and its BR-23 module
Proportion of patients with a change in fatigue condition | Change between baseline and 6 months and between 6 months and 12 months
  PFS-12 questionnaire
Proportion of patients with a change in health-related quality of life | Change between baseline and 6 months and between 6 months and 12 months
  EQ-5D-5L questionnaire
Proportion of patients who modify their professional status | Change between baseline and 6 months and between 6 months and 12 months
  Change in professional status, return to work, and perceived difficulty at work by a self-administered questionnaire.
Proportion of patients with a modification on serum circulating levels of endocrine factors (insulin, IGF1, estradiol) | Change between Day 0 and 6 months
  Blood sample
Proportion of patients with a modification on plasma circulating levels of cytokines (inflammatory cytokines: IL-6, TNF, and CRP; adipokines: adiponectin and leptin) | Change between Day 0 and 6 months
  Blood sample
Proportion of patients with a modification on vitamin D status | Change between Day 0 and 6 months
  Blood sample
Number of patients who accept the connected device | Baseline, 6 months and 12 months
  Self-administered qualitative questionnaire used in social psychology science
Number of patients who accept the therapeutic program | Baseline, 6 months and 12 months
  self-administered qualitative questionnaire used in social psychology science
Proportion of patients who refuse to participate | Baseline (day 0)
  Refusal rate among eligible patients to whom the study was presented

OTHER OUTCOMES:
Cost-utility of the interventions as assessed using clinical data (treatments received, patients' diary on medical consultations) and hospital costs (national data). | 12 months
  The cost-utility of implementing each intervention will be assessed.
Cost-effectiveness of the interventions as assessed using clinical data (treatments received, patients' diary on medical consultations), hospital costs (national data), and benefit in physical activity level. | 12 months
  The cost-effectiveness of implementing each intervention will be assessed.
Assessment of the association between the objective and subjective characteristics of living spaces and patients' PA practices. | 12 months
  ALPHA questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice Fervers, MD, PhD, Principal Investigator — Centre Léon Bérard, Lyon, France
Locations (3):
- France (3):
  - Institut Sainte-Catherine, Avignon
  - CHRU Besançon, Besançon
  - Centre Léon Bérard, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beasley JM, Kwan ML, Chen WY, Weltzien EK, Kroenke CH, Lu W, Nechuta SJ, Cadmus-Bertram L, Patterson RE, Sternfeld B, Shu XO, Pierce JP, Caan BJ. Meeting the physical activity guidelines and survival after breast cancer: findings from the after breast cancer pooling project. Breast Cancer Res Treat. 2012 Jan;131(2):637-43. doi: 10.1007/s10549-011-1770-1. Epub 2011 Sep 21. PMID 21935600
- [Background] Beg MS, Gupta A, Stewart T, Rethorst CD. Promise of Wearable Physical Activity Monitors in Oncology Practice. J Oncol Pract. 2017 Feb;13(2):82-89. doi: 10.1200/JOP.2016.016857. PMID 28387544
- [Background] Cadmus-Bertram LA, Marcus BH, Patterson RE, Parker BA, Morey BL. Randomized Trial of a Fitbit-Based Physical Activity Intervention for Women. Am J Prev Med. 2015 Sep;49(3):414-8. doi: 10.1016/j.amepre.2015.01.020. Epub 2015 Jun 10. PMID 26071863
- [Background] Ferguson T, Rowlands AV, Olds T, Maher C. The validity of consumer-level, activity monitors in healthy adults worn in free-living conditions: a cross-sectional study. Int J Behav Nutr Phys Act. 2015 Mar 27;12:42. doi: 10.1186/s12966-015-0201-9. PMID 25890168
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Ibrahim EM, Al-Homaidh A. Physical activity and survival after breast cancer diagnosis: meta-analysis of published studies. Med Oncol. 2011 Sep;28(3):753-65. doi: 10.1007/s12032-010-9536-x. Epub 2010 Apr 22. PMID 20411366
- [Background] Lahart IM, Metsios GS, Nevill AM, Carmichael AR. Physical activity, risk of death and recurrence in breast cancer survivors: A systematic review and meta-analysis of epidemiological studies. Acta Oncol. 2015 May;54(5):635-54. doi: 10.3109/0284186X.2014.998275. Epub 2015 Mar 9. PMID 25752971
- [Background] Sullivan AN, Lachman ME. Behavior Change with Fitness Technology in Sedentary Adults: A Review of the Evidence for Increasing Physical Activity. Front Public Health. 2017 Jan 11;4:289. doi: 10.3389/fpubh.2016.00289. eCollection 2016. PMID 28123997
- [Background] Thariat J, Creisson A, Chamignon B, Dejode M, Gastineau M, Hebert C, Boissin F, Topfer C, Gilbert E, Grondin B, Guennoc H, Mari V, Buzzo S, Saja D, Duboue N, Boulahssass R, Tosi A, Verne S, Ducray J, Benard-Thiery I, Ferrero JM. [Integrating patient education in your oncology practice]. Bull Cancer. 2016 Jul-Aug;103(7-8):674-90. doi: 10.1016/j.bulcan.2016.04.007. Epub 2016 Jun 7. French. PMID 27286758
- [Background] Tudor-Locke C, Hatano Y, Pangrazi RP, Kang M. Revisiting "how many steps are enough?". Med Sci Sports Exerc. 2008 Jul;40(7 Suppl):S537-43. doi: 10.1249/MSS.0b013e31817c7133. PMID 18562971
- [Derived] Touillaud M, Fournier B, Perol O, Delrieu L, Maire A, Belladame E, Perol D, Perrier L, Preau M, Leroy T, Fassier JB, Fillol F, Pascal S, Durand T, Fervers B. Connected device and therapeutic patient education to promote physical activity among women with localised breast cancer (DISCO trial): protocol for a multicentre 2x2 factorial randomised controlled trial. BMJ Open. 2021 Sep 13;11(9):e045448. doi: 10.1136/bmjopen-2020-045448. PMID 34518245